CLINICAL TRIAL: NCT05210699
Title: CSD201201: A Randomized, Open-Label, Crossover Study to Assess Elements of Abuse Liability for Electronic Nicotine Delivery System P12
Brief Title: CSD201201: Study to Assess Elements of Abuse Liability for Electronic Nicotine Delivery System P12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD201201
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product usage order A B N C E D (Experimental): Subjects will use each of the 5 products sequentially (A B N C E D) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product N
- Product usage order B C A D N E (Experimental): Subjects will use each of the 5 products sequentially (B C A D N E) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product N
- Product usage order C D B E A N (Experimental): Subjects will use each of the 5 products sequentially (C D B E A N) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product N
- Product usage order D E C N B A (Experimental): Subjects will use each of the 5 products sequentially (D E C N B A) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product N
- Product usage order E N D A C B (Experimental): Subjects will use each of the 5 products sequentially (E N D A C B) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product N
- Product usage order N A E B D C (Experimental): Subjects will use each of the 5 products sequentially (N A E B D C) during an evaluation period, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product N

INTERVENTIONS:
Other: Product A — Usual Brand (UB) filtered, menthol combustible cigarette
Other: Product B — Flavor variant P1211216 of a 1.5% nicotine ENDS product
Other: Product C — Flavor variant P1211217 of a 2.4% nicotine ENDS product
Other: Product D — Flavor variant P1211222 of a 5.0% nicotine ENDS product
Other: Product E — Flavor variant P1213616 of a 1.5% nicotine ENDS product
Other: Product N — Nicorette® White Ice Mint 4 mg nicotine gum

SUMMARY:
This is a randomized, open-label, 6-way crossover, multi-site study designed to evaluate elements of abuse liability (AL) including subjective effects and physiological measures (pharmacodynamics [PD]), and nicotine uptake (pharmacokinetics [PK]) during and following ad libitum use of the Electronic Nicotine Delivery Systems (ENDS) investigational products (IPs) in generally healthy combustible cigarette (CC) smokers and dual users of CC and ENDS.

DETAILED DESCRIPTION:
The study will evaluate elements of AL of ENDS IPs against CC and nicotine polacrilex gum in generally healthy menthol CC smokers of and dual users of CC and ENDS in a confinement setting.

Potential subjects will complete a pre-screening interview and a Screening Visit to assess eligibility within 45 days prior to enrollment, randomization and confinement.

Starting on Study Day 1, eligible subjects will be randomized to 1 of 6 IP use sequences (based on a Williams Design) and will be confined at the clinical site for 8 days and 7 nights to complete the study.

On Day 3 and continuing through Day 8, subjects in each arm will participate in six separate Test Sessions, one for each IP, that will last for approximately 4 hours following the start of IP use. During each Test Session, subjects will use one of the six IPs: four ENDS IPs, a high-AL comparator (subject's UB cigarette) and a low-AL comparator (a commercially available nicotine gum for nicotine replacement therapy), based on the assigned IP use sequences. ENDS IP cartridges will be weighed prior to and after product use in the Test Session. Each Test Session will include collection of both PD measures (subjective and physiological) and PK measures prior to, during, and following IP use.

Subjects will acclimate to the assigned products prior to each Test Session. On Study Day 1 (Pre-study Product Acclimation Period), subjects will use each of five IPs (four ENDS IPs and one nicotine gum) at least once. In addition, on the half day prior to each respective Test Session (Starting on Day 2), subjects will participate in a Product Acclimation Period in which they will use the randomized IP (to be tested during the following day's Test Session, to include ENDS or nicotine gum) at least four times . Subjects will have access to UB cigarette for ad libitum use at any time during Pre-Study Product Acclimation period and Product Acclimation Periods as long as they meet the IP acclimation criteria. At the end of each Product Acclimation Period, there will be a required 12-hour abstinence period from use of tobacco/nicotine containing products prior to the Test Session the following day. The study will complete when all six IPs have been tested.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Expired breath carbon monoxide level is ≥ 10 ppm and ≤ 100 ppm at Screening.
4. Positive urine cotinine test at Screening.
5. Smokes only combustible, filtered, menthol cigarettes, 83 mm to 100 mm in length.
6. Agrees to smoke same usual brand (UB) cigarette throughout the study period. UB cigarette is defined as the cigarette brand style currently smoked most frequently by the subject.
7. Subjects must meet one (a or b) of the following tobacco use conditions:

   1. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Principal Investigator (PI).
   2. Dual user of combustible cigarettes and electronic cigarettes (ECs) who self-reports:

   i. Smoking at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening Visit. Brief periods of abstinence more than 30 days prior to screening due to illness, quit attempt or clinical study participation will be allowed at the discretion of the Investigator and ii. Using a nicotine-containing ENDS (cartridge or a tank system).
8. Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes."
9. Willing to use UB cigarette, ENDS, and Nicorette gum during the study period.
10. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each Test Session.
11. Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until End-of-Study.
12. Agrees to in-clinic confinement of 8 days and 7 nights.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at Screening and at check-in Day 1.
4. Weight of ≤ 110 pounds.
5. Hemoglobin level is < 12.5 for females or <13.0 for males g/dL at Screening.
6. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
9. Must not be a current regular user (i.e., > 5 times per month) of any tobacco products other than CCs or ENDS within the last 6 months prior to screening.
10. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
11. History or presence of bleeding or clotting disorders.
12. Any use of anticoagulants or daily use of aspirin (≥ 325 mg).
13. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent and between Screening and check-in Day 1.
14. Plasma donation within (≤) 7 days prior to the signing of informed consent and between Screening and check-in Day 1.
15. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
16. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
17. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
18. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Day 1.
19. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous quit attempt within (≤) 30 days prior to the signing of the ICF.
20. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol breathalyzer result at Screening or Day 1.
21. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
AUECPL 3-240 | 5 minutes to 240 minutes
  area-under-the-effects curve (AUEC) for product liking (PL) numeric rating scale (NRS) score-versus-time curve from 3 minutes to 240 minutes after the start of IP use. Product Liking is a numeric rating scale ranging from 0 to 10. A higher score indicates a higher liking of the product.
Emax PL | 240 minutes
  maximum product liking (PL) numeric rating scale (NRS) score after the start of IP use. Product Liking is a numeric rating scale ranging from 0 to 10. A higher score indicates a higher liking of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hong, MD, Study Director — RAIS
Locations (2):
- United States (2):
  - QPS Bio-Kinetic, Springfield, Missouri
  - AMR Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No